CLINICAL TRIAL: NCT05604144
Title: A Proof-of-Concept Study to Define the Safety, Efficacy and Feasibility of Cryoanalgesia (Iovera°®) for the Treatment of Pain in Subjects With Morton's Neuroma
Brief Title: Cryoanalgesia for the Treatment of Pain in Subjects With Morton's Neuroma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northern California Research Trials, Inc. (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry); NorthBay Healthcare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IITMN001
Record Dates: First submitted 2022-10-04; First posted 2022-11-03 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Morton's Neuroma; Pain Management
Keywords: Proof-of-Concept; Pilot Study; Podiatric Pain Management; Cryoanalgesia
MeSH Terms: conditions — Morton Neuroma; Agnosia

STUDY DESIGN:
Intervention Model Description: Proof-of-Concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active Treatment (Other): As a Proof of Concept Study, 5 subjects will follow the same protocol, with one cryoanalgesic treatment (iovera°®) with a 6 month clinical follow-up.
  Interventions: Device: Cryoanalgesia (iovera°®)

INTERVENTIONS:
Device: Cryoanalgesia (iovera°®) — iovera°® treatment will be administered via ultrasound guidance to 1-2 branches of the dorsal/digital/proper nerve/s that innervate the Morton's neuroma. The treatment will be completed one time per subject.
  Other Names: iovera°®

SUMMARY:
This is a Proof-of-Concept Trial to define the safety, efficacy and feasibility of a cryoanalgesic device (iovera°®) for the treatment of pain in subjects diagnosed with Morton's Neuroma, who have failed conservative therapies.

DETAILED DESCRIPTION:
Hypothesis:

Cryoanalgesia (iovera°®) will provide a safe, effective and feasible tool as a pain medicine modality to offer analgesic pain relief in patients with Morton's Neuroma, thereby introducing a new non-opioid therapeutic option to these patients in need.

Primary Objective:

To define and characterize the analgesic effect following a single cryoanalgesic application to the Dorsal, Digital Proper Nerve/s in subjects diagnosed with Morton's Neuroma, who have failed conservative therapies.

Primary Endpoints:

1. The area under the curve of the Numeric Rating Scale (NRS) Pain Intensity Scores; the NRS is a 0 to 10 rating scale with the number "0" indicating "no pain" and the number "10" indicating the "worst possible pain". The NRS is completed by subjects three times per day from Day 0 to 3 months post treatment, then the NRS will be done weekly through 6 months post treatment. 2. The total daily opioid consumption will be evaluated from Day 0 to 6 months post treatment to determine if the cryoanalgesic treatment decreased the subject's daily opioid pain management requirement.

Secondary Objectives:

1. Safety: To define the incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) related to treatment.
2. Efficacy: To assess the cryoanalgesic application as defined by both the subject and physician; to define the impact of treatment related to ambulatory steps pre and post procedure.
3. Feasibility: To characterize and compare the cryoanalgesic treatment process to Standard of Care (SOC) treatment modalities.

Secondary Endpoints:

1. Safety Endpoints: The incidence of treatment emergent AEs and SAEs will be recorded and evaluated from the date of the cryoanalgesic application through 6 months post treatment.
2. Efficacy Endpoints: Ambulatory steps/distance will be recorded during the Screening Period and through 90 days post treatment. A wrist device will track the subjects daily steps (ambulation) before and after the cryoanalgesic treatment. Tracking the subject's daily steps before and after treatment may offer an objective measure of cryoanalgesic efficacy. Both Subject and Physician Satisfaction Questionnaires will be recorded from Day 0 post-treatment through the following 6 months. These standardized questionnaires describe how satisfied or unsatisfied the subjects and physician are from the cryoanalgesic treatment.
3. Feasibility Endpoints: Physician Feasibility Questionnaires will define treatment approaches, device utilization and impact on the subject's clinical course compared to Standard of Care treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers ages 18 or older.
2. Able to provide informed consent, adhere to the study schedule, and complete all study assessments.
3. Body Mass Index (BMI) ≥18 and ≤40 kg/m2.
4. Unilateral Morton's Neuroma diagnosed by MRI.
5. Subject has failed conservative treatment options.

Exclusion Criteria:

1. Documented allergy, hypersensitivity, intolerance, or contraindication to amide-type local anesthetics (i.e., lidocaine), or opioids, NSAIDs.
2. Documented history of uncontrolled diabetes, bleeding disorder, severe Peripheral Vascular Disease (PVD).
3. Concurrent painful physical condition that may require analgesic treatment (i.e., long-term opioid use) which, in the Principal Investigator's opinion, may confound the treatment assessments.
4. History of, suspected, or known addiction to/or abuse of illicit drug/s, prescription medicine/s, or alcohol within the past 3 years.
5. Administration of an investigational drug or medical device within 30 days of the Screening Period.
6. Previous participation in a cryoneurolysis study.
7. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Principal Investigator, could potentially interfere with study assessments or compliance.
8. Currently pregnant, nursing, or planning to become pregnant during the study.
9. Clinically significant medical disease that, in the opinion of the Principal Investigator, would make participation in a clinical study inappropriate.
10. Inadequate sensory function of the affected foot (as defined at the Screening Visit Neurologic Lower Extremity (LE) exams).
11. Any clinically significant event or condition uncovered during the Screening Period (e.g., contra-lateral foot injury) that, in the opinion of the Principal Investigator, renders the subject medically unstable or complicates the subject's study participation.
12. Subject has a history of: Cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria or Raynaud's Disease.
13. Subject has an active, wound, open and/or potential infection near the anticipated treatment site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-04-22 (Estimated); Study Completion 2023-04-22 (Estimated)

PRIMARY OUTCOMES:
Pain Management | Six Months
  Numeric Rating Scale (NRS) Pain Intensity Scores completed by subjects three times per day from Day 0 to 3 months post treatment, then NRS weekly through 6 months post treatment. 2. The total daily opioid consumption from Day 0 to 6 months post treatment.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | Six Months
  The incidence of treatment emergent AEs and SAEs will be recorded and evaluated from the date of the treatment through 6 months post treatment.
Ambulation | Six Months
  Ambulatory steps/distance will be recorded during the Screening Period and through 90 days post treatment. Both Subject and Physician Satisfaction Questionnaires will be recorded from Day 0 post-treatment through the following 6 months.
Medical Device Feasibility | Six Months
  Physician Feasibility Questionnaires will define treatment approaches, device utilization and impact on the subject's clinical course compared to SOC treatment modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Miller, DPM, FACPM, FFPM, Principal Investigator — NorthBay Healthcare
Locations (2):
- United States (2):
  - NorthBay Healthcare, Fairfield, California
  - NorthBay Healthcare, Vacaville, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cleveland Clinic Communication: Morton's Neuroma: Causes, Symptoms, Diagnois & Treatment. https://my.cleveland clinic.org/health/diseases/15118-mortons-neuroma pages 1-13.
- [Background] Matthews BG, Hurn SE, Harding MP, Henry RA, Ware RS. The effectiveness of non-surgical interventions for common plantar digital compressive neuropathy (Morton's neuroma): a systematic review and meta-analysis. J Foot Ankle Res. 2019 Feb 13;12:12. doi: 10.1186/s13047-019-0320-7. eCollection 2019. PMID 30809275
- [Background] Sidon E, Rogero R, McDonald E, Daecher A, Shakked R, Pedowitz DI, Fuchs D, Daniel JN, Raikin SM. Prevalence of Neuropathic Pain Symptoms in Foot and Ankle Patients. Foot Ankle Int. 2019 Jun;40(6):629-633. doi: 10.1177/1071100719838302. Epub 2019 Mar 22. PMID 30902025
- [Background] Thomson L, Aujla RS, Divall P, Bhatia M. Non-surgical treatments for Morton's neuroma: A systematic review. Foot Ankle Surg. 2020 Oct;26(7):736-743. doi: 10.1016/j.fas.2019.09.009. Epub 2019 Nov 2. PMID 31718949
- [Background] Ferkel E, Davis WH, Ellington JK. Entrapment Neuropathies of the Foot and Ankle. Clin Sports Med. 2015 Oct;34(4):791-801. doi: 10.1016/j.csm.2015.06.002. PMID 26409596
- [Background] Ross AB, Jacobs A, Williams KL, Bour RK, Gyftopoulos S. Ultrasound-Guided Injection Treatments Versus Surgical Neurectomy for Morton Neuroma: A Cost-Effectiveness Analysis. AJR Am J Roentgenol. 2022 Feb;218(2):234-240. doi: 10.2214/AJR.21.26419. Epub 2021 Sep 15. PMID 34523955
- [Background] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Background] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Background] Davis T, Loudermilk E, DePalma M, Hunter C, Lindley D, Patel N, Choi D, Soloman M, Gupta A, Desai M, Buvanendran A, Kapural L. Prospective, Multicenter, Randomized, Crossover Clinical Trial Comparing the Safety and Effectiveness of Cooled Radiofrequency Ablation With Corticosteroid Injection in the Management of Knee Pain From Osteoarthritis. Reg Anesth Pain Med. 2018 Jan;43(1):84-91. doi: 10.1097/AAP.0000000000000690. PMID 29095245
- [Background] Poppler LH, Parikh RP, Bichanich MJ, Rebehn K, Bettlach CR, Mackinnon SE, Moore AM. Surgical interventions for the treatment of painful neuroma: a comparative meta-analysis. Pain. 2018 Feb;159(2):214-223. doi: 10.1097/j.pain.0000000000001101. PMID 29189515